CLINICAL TRIAL: NCT03035370
Title: A Phase I Dose Escalation Randomized, Double-blind, Placebo-controlled Safety and Immunogenicity Trial of the Reactivation of Pertussis Toxin Immunity With the Viaskin Epicutaneous Delivery System in Healthy Adults
Brief Title: Viaskin Pertussis Vaccine Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: DBV Technologies (Industry)
Collaborators: University Hospital, Geneva (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: VBEST
Record Dates: First submitted 2016-03-15; First posted 2017-01-30 (Estimated); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Whooping Cough
Keywords: Pertussis; Epicutaneous ImmunoTherapy (EPIT); Vaccine; Viaskin PT
MeSH Terms: conditions — Whooping Cough | interventions — Boostrix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Viaskin PT 25 mcg (Experimental): Viaskin PT 25 mcg
  Interventions: Biological: Viaskin PT 25 mcg; Biological: Boostrix™
- Viaskin PT 50 mcg (Experimental): Viaskin PT 50 mcg
  Interventions: Biological: Viaskin PT 50 mcg; Biological: Boostrix™
- Viaskin PT Placebo (Placebo Comparator): Viaskin PT Placebo
  Interventions: Biological: Viaskin PT Placebo; Biological: Boostrix™

INTERVENTIONS:
Biological: Viaskin PT 25 mcg — Two applications of Viaskin 25 mcg PT at a 2-week interval (D0 and D14).
  Arms: Viaskin PT 25 mcg
Biological: Viaskin PT 50 mcg — Two applications of Viaskin 50 mcg PT at a 2-week interval (D0 and D14).
  Arms: Viaskin PT 50 mcg
Biological: Viaskin PT Placebo — Two applications of Viaskin PT Placebo at a 2-week interval (D0 and D14).
  Arms: Viaskin PT Placebo
Biological: Boostrix™ — Four weeks after the second Viaskin application (at Day 42 of the study), all subjects will receive a dose of diphtheria-tetanus-pertussis vaccine (Boostrix® dTpa) to ensure the optimal recall of their immunity against pertussis.

SUMMARY:
The study is a Phase I, first in human, monocenter study, aiming at assessing the safety and immunogenicity of a genetically detoxified pertussis toxin (PT) when administered via the cutaneous route with Viaskin patches to healthy volunteers at 2 different doses of 25 mcg or 50 mcg PT protein compared to Viaskin placebo.

Two cohorts of 30 subjects will be successively enrolled. Safety of the product will be assessed throughout the 10-week study and its immunogenicity will be assessed at regular intervals with collection of blood samples for immunological analyses.

Four weeks after the second Viaskin application (at Day 42 of the study), all subjects will receive a dose of diphtheria-tetanus-pertussis vaccine (Boostrix® dTpa) to ensure the optimal recall of their immunity against pertussis.

ELIGIBILITY:
Inclusion Criteria:

* Has provided written informed consent before enrollment;
* Adult male or female, ages 18 to 40 years (inclusive) at the time of enrollment;
* Non-pregnant, non-lactating female;
* Free of clinically significant health problems, as determined by pertinent medical history and clinical examination at study screening;
* With documented history of pertussis immunization (at least 4 doses);
* Women of childbearing potential with a negative pregnancy test at entry;
* Females of childbearing potential who are willing to use an effective method of contraception.

Exclusion Criteria:

* Prior dTpa immunization within the last 10 years or prior dT immunization within the last 2 years, or any other investigational vaccine likely to impact on interpretation of the trial data;
* Suspected or confirmed pertussis infection within the last 10 years or documented pertussis infection in a household member within the last 10 years;
* Receipt of licensed vaccines within 14 days of planned study immunization (30 days for live vaccines) or ongoing participation in another clinical interventional trial.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2016-09-05 (Actual); Primary Completion 2018-04-25 (Actual); Study Completion 2018-04-25 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (AE). | From Day 0 to Day 70.
  * Solicited AEs occurring from the time of each application through 14 days following Viaskin PT application;
  * Unsolicited AEs from the time of application through 28 days following the 1st application;
  * Serious Adverse Events from the time of the inform consent form signature through the final study visit of subject.

SECONDARY OUTCOMES:
PT-specific antibody response (anti-PT IgG antibodies and PT-specific neutralizing antibodies). | Day 14, Day 28, Day 42, Day 70.

CONTACTS AND LOCATIONS:
Overall Officials: Claire Anne Siegrist, M.D, Principal Investigator — Medical Faculty (UNIGE) and University hospital of Geneva , Center of Vaccinology
Locations (1):
- Center for Vaccinology Medical faculty UNIGE and University of Geneva (HUG), Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Chatzis O, Blanchard-Rohner G, Mondoulet L, Pelletier B, De Gea-Hominal A, Roux M, Huttner A, Herve PL, Rohr M, Matthey A, Gutknecht G, Lemaitre B, Hayem C, Pham HT, Wijagkanalan W, Lambert PH, Benhamou PH, Siegrist CA. Safety and immunogenicity of the epicutaneous reactivation of pertussis toxin immunity in healthy adults: a phase I, randomized, double-blind, placebo-controlled trial. Clin Microbiol Infect. 2021 Jun;27(6):878-885. doi: 10.1016/j.cmi.2020.08.033. Epub 2020 Sep 5. PMID 32896653